CLINICAL TRIAL: NCT06293365
Title: A Randomized, Two-period Crossover Study to Demonstrate the Comparability of Pharmacokinetics of Subcutaneous Ianalumab Between 2mL Auto-injector/2mL Pre-filled Syringe With 1 mL Pre-filled Syringe in Adult Participants With Autoimmune Disease
Brief Title: Two-period Crossover Study to Demonstrate the Comparability of Pharmacokinetics of Subcutaneous Ianalumab Between 2mL Auto-injector/2mL PFS with1mL Pre-filled Syringe in Adult Participants With Autoimmune Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CVAY736A2202; 2023-508996-35-00 (Registry Identifier: EU CT NUMBER)
Expanded Access: NCT07244289 (Available)
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Sjögrens Disease; Systemic Lupus Erythematosus; Rheumatoid Arthritis
Keywords: Sjögrens Disease (SjD); Systemic lupus erythematosus (SLE); Rheumatoid Arthritis (RA); Pharmacokinetic (PK) comparability; 2 mL auto-injector (AI); 1 mL pre-filled syringe (PFS); 2 mL pre-filled syringe (PFS); VAY736; ianalumab; B cell depletion; Area under the curve (AUC); Cmax
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis, Rheumatoid | interventions — ianalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Cohort 1: Sequence 1 + Thigh (Experimental): Patients randomized to receive injection (2 x 1 mL) PFS in TP1 in Thigh (1 X 2 mL) AI in TP2 in Thigh
  (1 x 2 mL) AI in ETP in Thigh/ Abdomen
  Interventions: Biological: VAY736 1ml PFS; Biological: VAY736 2ml AI
- Cohort 1: Sequence 1 + Abdomen (Experimental): Patients randomized to receive injection
  1. X 2 mL) AI in TP1 in Abdomen
  2. x 1 mL) PFS in TP2 in Abdomen
  (1 x 2 mL) AI in ETP in Thigh/ Abdomen
  Interventions: Biological: VAY736 1ml PFS; Biological: VAY736 2ml AI
- Cohort 1: Sequence 2 + Thigh (Experimental): Patients randomized to receive injection (2 x 1 mL) PFS in TP1 in Thigh (1 X 2 mL) AI in TP2 in Thigh
  (1 x 2 mL) AI in ETP in Thigh/ Abdomen
  Interventions: Biological: VAY736 1ml PFS; Biological: VAY736 2ml AI
- Cohort 1: Sequence 2 + Abdomen (Experimental): Patients randomized to receive injection
  1. X 2 mL) AI in TP1 in Abdomen
  2. x 1 mL) PFS in TP2 in Abdomen
  (1 x 2 mL) AI in ETP in Thigh/ Abdomen
  Interventions: Biological: VAY736 1ml PFS; Biological: VAY736 2ml AI
- Cohort 2: Sequence 1 + Thigh (Experimental): Patients randomized to receive injection (2 x 1 mL) PFS in TP1 in Thigh
  1. X 2 mL) PFS in TP2 in Thigh
  2. x 1 mL) PFS in ETP in Thigh/ Abdomen/ Upper Arm
  Interventions: Biological: VAY736 1ml PFS; Biological: VAY736 2 ml PFS
- Cohort 2: Sequence 1 + Abdomen (Experimental): Patients randomized to receive injection
  1. X 2 mL) PFS in TP1 in Abdomen
  2. x 1 mL) PFS in TP2 in Abdomen
  (2 x 1 mL) PFS in ETP in Thigh/ Abdomen/ Upper Arm
  Interventions: Biological: VAY736 1ml PFS; Biological: VAY736 2 ml PFS
- Cohort 2: Sequence 1 + Upper Arm (Experimental): Patients randomized to receive injection (2 x 1 mL) PFS in TP1 in Upper Arm
  1. X 2 mL) PFS in TP2 in Upper Arm
  2. x 1 mL) PFS in ETP in Thigh/ Abdomen/ Upper Arm
  Interventions: Biological: VAY736 1ml PFS; Biological: VAY736 2 ml PFS
- Cohort 2: Sequence 2 + Thigh (Experimental): Patients randomized to receive injection
  1. X 2 mL) PFS in TP1 in Thigh
  2. x 1 mL) PFS in TP2 in Thigh
  (2 x 1 mL) PFS in ETP in Thigh/ Abdomen/ Upper Arm
  Interventions: Biological: VAY736 1ml PFS; Biological: VAY736 2 ml PFS
- Cohort 2: Sequence 2 + Abdomen (Experimental): Patients randomized to receive injection (2 x 1 mL) PFS in TP1 in Abdomen
  1. X 2 mL) PFS in TP2 in Abdomen
  2. x 1 mL) PFS in ETP in Thigh/ Abdomen/ Upper Arm
  Interventions: Biological: VAY736 1ml PFS; Biological: VAY736 2 ml PFS
- Cohort 2: Sequence 2 + Upper Arm (Experimental): Patients randomized to receive injection
  1. X 2 mL) PFS in TP1 in Upper Arm
  2. x 1 mL) PFS in TP2 in Upper Arm
  (2 x 1 mL) PFS in ETP in Thigh/ Abdomen/ Upper Arm
  Interventions: Biological: VAY736 1ml PFS; Biological: VAY736 2 ml PFS

INTERVENTIONS:
Biological: VAY736 1ml PFS — Solution for injection.
  Other Names: Ianalumab
Biological: VAY736 2 ml PFS — Solution for injection
  Other Names: Ianalumab
  Arms: Cohort 2: Sequence 1 + Abdomen; Cohort 2: Sequence 1 + Thigh; Cohort 2: Sequence 1 + Upper Arm; Cohort 2: Sequence 2 + Abdomen; Cohort 2: Sequence 2 + Thigh; Cohort 2: Sequence 2 + Upper Arm
Biological: VAY736 2ml AI — Solution for injection.
  Other Names: Ianalumab
  Arms: Cohort 1: Sequence 1 + Abdomen; Cohort 1: Sequence 1 + Thigh; Cohort 1: Sequence 2 + Abdomen; Cohort 1: Sequence 2 + Thigh

SUMMARY:
The purpose of this study is to demonstrate the comparability of ianalumab exposure following the sub-cutaneous (s.c.) administration of one injection of 300 mg/2 mL auto-injector (AI) versus two injections of 150 mg/1 mL pre-filled syringe (PFS), and to evaluate the safety and tolerability of ianalumab following the s.c. administration of both devices in participants with rheumatoid arthritis (RA), Sjögren's disease (SjD), or systemic lupus erythematosus (SLE).

A second cohort will be included with the objective of demonstrating the comparability of pharmacokinetics of ianalumab between 1 x 2 mL Pre-filled Syringe (PFS) and 2 x 1 mL PFS.

DETAILED DESCRIPTION:
The study consists of the following periods:

Screening period (up to 4 weeks):

Following the signing of the informed consent, participants will be assessed for eligibility during this period of up to 4 weeks.

Treatment Period 1 + Treatment Period 2, (Week 0 to Week 24):

After completion of the screening period, eligible participants will be randomized at the Baseline visit (Week 0) to one of the 2 treatment sequences (treatment switch at Week 12) in a ratio of 1:1 described below:

* Cohort 1:

  * Sequence 1: ianalumab 300 mg s.c. (2 x 1 mL PFS) monthly + SoC in Treatment Period 1 and ianalumab 300 mg s.c. (1 x 2 mL AI) monthly + SoC in Treatment Period 2
  * Sequence 2: ianalumab 300 mg s.c. (1 x 2 mL AI) monthly + SoC in Treatment Period 1 and ianalumab 300 mg s.c. (2 x 1 mL PFS) monthly + SoC in Treatment Period 2
* Cohort 2:

  * Sequence 1: ianalumab 300 mg s.c. (2 x 1 mL PFS) monthly + SoC in Treatment Period 1 and ianalumab 300 mg s.c. (1 x 2 mL PFS) monthly + SoC in Treatment Period 2
  * Sequence 2: ianalumab 300 mg s.c. (1 x 2 mL PFS) monthly + SoC in Treatment Period 1 and ianalumab 300 mg s.c. (2 x 1 mL PFS) monthly + SoC in Treatment Period 2 In addition, within each sequence, participants will be further randomized to one of the predetermined injection sites with equal allocation, resulting in a total randomization combination of four (2 sequences x 2 injection sites) for Cohort 1 and six (2 sequences x 3 injection sites) for Cohort 2, respectively.

Extended Treatment period (Week 24 to Week 72): After completion of Week 24 assessment, all participants (who did not discontinue during treatment period) will have the option to enter the extended treatment period to receive ianalumab 300 mg s.c. (Cohort 1: 2 mL AI; Cohort 2: 2 x 1 mL PFS) monthly up to Week 68. The end of treatment (EOT) visit will be performed 4 weeks after the last study treatment administration, i.e., at Week 72.

Mandatory Post-Treatment safety follow-up period (from Week 72 to Week 88): Participants who completed the last study treatment or prematurely discontinued from study treatment will enter the post-treatment safety follow-up period.

Conditional Post-Treatment safety follow-up period (from Week 88 to Week 176) Post-treatment follow-up will be performed until B-cell recovery or up to 2 years. B-cell recovery is defined when CD19+ B-cell counts return to >= 50 cells/μL or >= 80% of baseline value, whichever occurs earlier.

ELIGIBILITY:
Key Inclusion criteria:

* Signed informed consent must be obtained before any assessment is performed.
* Male and female patients aged 18 years to 70 years (inclusive).
* Body weight at least 35 kg and not more than 150 kg and must have a body mass index (BMI) within the range of 18 - 35 kg/m2. BMI = Body weight (kg) / [Height (m)]2 at screening.
* Diagnosed with RA, SjD and/or SLE as determined by the investigator.
* Have active disease (RA, SjD or SLE) that may benefit from B-cell depletion therapy, as determined by the investigator.
* Participants currently receiving protocol-allowed SoC should be on stable doses of SoC medications for 4 weeks prior to first dosing of study treatment.
* Ability to communicate well with the investigator, understand and agree to comply with the requirements of the study.

Key Exclusion criteria:

* Use of prohibited therapies.
* Active viral, bacterial or other infections requiring systemic treatment at the time of screening or baseline or history of recurrent clinically significant infection.
* Plans for administration of live vaccines during the study period.
* Uncontrolled co-existing serious disease.
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, refusing or unable to use highly effective methods of contraception while on study treatment and for 6 months after stopping of study drug.
* US (and other countries, if locally required): sexually active males unless using barrier protection during intercourse with women of child-bearing potential while taking study treatment.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2029-01-04 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Area under the curve (AUC) calculated to the end of a dosing interval (tau) at steady-state (AUCtau) for ianalumab | Over a dosing interval after 3rd (between Week 8 and 12) and 6th dose (between Week 20 and 24).
  To demonstrate the pharmacokinetics (PK) comparability of ianalumab 300 mg s.c. at steady state between the 1 x 2 mL AI and 2 x 1 mL PFS
Cohort 1: Maximum (peak) observed serum drug concentration after dose administration (Cmax) for ianalumab | Over a dosing interval after 3rd (between Week 8 and 12) and 6th dose (between Week 20 and 24).
  To demonstrate the pharmacokinetics (PK) comparability of ianalumab 300 mg s.c. at steady state between the 1 x 2 mL AI and 2 x 1 mL PFS
Cohort 2: Area under the curve (AUC) calculated to the end of a dosing interval (tau) at steady-state (AUCtau) for ianalumab | Over a dosing interval after 3rd (between Week 8 and 12) and 6th dose (between Week 20 and 24).
  To demonstrate the pharmacokinetics (PK) comparability of ianalumab 300 mg s.c. at steady state between the 1 x 2 mL PFS and 2 x 1 mL PFS.
Cohort 2: Maximum (peak) observed serum drug concentration after dose administration (Cmax) for ianalumab | Over a dosing interval after 3rd (between Week 8 and 12) and 6th dose (between Week 20 and 24).
  To demonstrate the pharmacokinetics (PK) comparability of ianalumab 300 mg s.c. at steady state between the 1 x 2 mL PFS and 2 x 1 mL PFS.

SECONDARY OUTCOMES:
Cohort 1: Time to reach maximum (peak) serum drug concentration following dose administration (Tmax) for ianalumab | After the 3rd and 6th dose
  To evaluate the pharmacokinetics of ianalumab 300 mg s.c. at steady state under the 1 x 2 mL AI and 2 x 1 mL PFS
Cohort 2: Time to reach maximum (peak) serum drug concentration following dose administration (Tmax) for ianalumab | After the 3rd and 6th dose
  To evaluate the pharmacokinetics of ianalumab 300 mg s.c. at steady state under the 1 x 2 mL PFS and 2 x 1 mL PFS
Cohort 1: Concentration at the end of a dosing interval (Ctrough) for ianalumab | At the end of dosing interval
  To evaluate the pharmacokinetics of ianalumab 300 mg s.c. at steady state under the 1 x 2 mL AI and 2 x 1 mL PFS
Cohort 2: Concentration at the end of a dosing interval (Ctrough) for ianalumab | At the end of dosing interval
  To evaluate the pharmacokinetics of ianalumab 300 mg s.c. at steady state under the 1 x 2 mL PFS and 2 x 1 mL PFS
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From date of randomization until 30 days safety follow-up, assessed up to approximately 56 months
  To evaluate the safety and tolerability of ianalumab administered 300 mg s.c. monthly.
Anti-ianalumab antibodies (ADA) | From date of randomization until 30 days safety follow-up, assessed up to approximately 56 months
  To assess the immunogenicity of ianalumab administered 300 mg s.c. monthly
Incidence of ADA positive participants | From date of randomization until 30 days safety follow-up, assessed up to approximately 56 months
  To assess the immunogenicity of ianalumab administered 300 mg s.c. monthly

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (35):
- United States (17):
  - Pinnacle Research Group Llc, Anniston, Alabama
  - Providence Medical Foundation, Fullerton, California
  - Advanced Medical Research, La Palma, California
  - Conquest Research, Winter Park, Florida
  - Parris and Associates Rheumatology, Lawrenceville, Georgia
  - Indiana Univ School of Dentistry, Indianapolis, Indiana
  - Ochsner Health System, Baton Rouge, Louisiana
  - Ahmed Arif Medical Research Center, Grand Blanc, Michigan
  - Paramount Med Rsrch and Consult LLC, Middleburg Heights, Ohio
  - RAO Research LLC, Oklahoma City, Oklahoma
  - Altoona Center for Clin Res, Duncansville, Pennsylvania
  - West Tennessee Research Institute, Jackson, Tennessee
  - Shelby Research LLC, Memphis, Tennessee
  - Novel Research LLC, Bellaire, Texas
  - Southwest Rheum Rsrch LLC, Mesquite, Texas
  - Uni of Texas Health Science Center, San Antonio, Texas
  - Advanced Rheumatology of Houston, Spring, Texas
- Argentina (3):
  - Novartis Investigative Site, Quilmes, Buenos Aires
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
- Canada (4):
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Rimouski, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Czechia (3):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Uherské Hradiště
- Hungary (2):
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Budapest
- Novartis Investigative Site, Salerno, SA, Italy
- Poland (2):
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lublin
- Spain (3):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com